CLINICAL TRIAL: NCT01842308
Title: A Phase 1/2 Trial of Carfilzomib and Melphalan and Conditioning for Autologous Stem Cell Transplantation for Multiple Myeloma (CARAMEL)
Brief Title: Carfilzomib and Melphalan Before Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1185; NCI-2013-00550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1185 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2019-10

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): CONDITIONING: Patients receive carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive melphalan IV over 1 hour on days -4 and -3.
  TRANSPLANT: Patients undergo autologous stem cell transplant on day 0.
  Interventions: Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carfilzomib; Other: Laboratory Biomarker Analysis; Drug: Melphalan

INTERVENTIONS:
Procedure: Autologous Bone Marrow Transplantation — Undergo autologous stem cell transplant
  Other Names: ABMT; Autologous Bone Marrow Transplant; Autologous Marrow Transplantation
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplantation
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813

SUMMARY:
This phase I/II trial studies the side effects and best dose of carfilzomib when given together with melphalan and to see how well they work in treating patients with multiple myeloma before stem cell transplant. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving carfilzomib together with melphalan may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of carfilzomib that can be added to high dose melphalan as part of conditioning chemotherapy for myeloma. (Phase I) II. To determine the efficacy of the combination in patients with myeloma undergoing stem cell transplantation, as defined by achievement of complete response (CR). (Phase II)

SECONDARY OBJECTIVES:

I. To examine the toxicities associated with addition of carfilzomib to high dose melphalan in patients with multiple myeloma (MM).

II. To determine the progression free rate at 1 and 2 years post registration.

TERTIARY OBJECTIVES:

I. To determine the proportion of patients achieving a minimal residual disease (MRD) negative status.

II. To assess the HevyLite assay prior to and during treatment.

OUTLINE: This is a phase I, dose-escalation study of carfilzomib followed by a phase II study.

CONDITIONING: Patients receive carfilzomib intravenously (IV) over 30 minutes on days -6, -5, -2, and -1. Patients also receive melphalan IV over 1 hour on days -4 and -3.

TRANSPLANT: Patients undergo autologous stem cell transplant on day 0.

After completion of study treatment, patients are followed up at day 30, day 100, and then every 90 days for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine =< 2 mg/dL
* Absolute neutrophil count >= 1000/uL
* Platelet count >= 50,000/uL
* Hemoglobin >= 8.0 g/dL
* Diagnosis of symptomatic MM
* Measurable disease of multiple myeloma at the time of baseline values for disease assessment as defined by at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >=10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Bone marrow plasma cells >= 30%
  * NOTE: For patients with no relapse prior to transplant, measurable disease at the time of diagnosis
  * NOTE: For patients who have had a disease relapse prior to transplant, measurable disease at the time of the most recent relapse immediately prior to transplant; NOTE: If the patient had treatment for the relapsed disease prior to transplant, the patient must have measurable disease at the time of relapse prior to this therapy
* Patient is considered for autologous stem cell transplantation with full dose melphalan (200 mg/m^2)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Recovered from toxicity of previous chemotherapy (excludes grade 1 neurotoxicity and hematological toxicity)
* Provide informed written consent
* Ejection fraction >= 45%
* Corrected pulmonary diffusion capacity of greater than or equal to 50%
* Forced expiratory volume in 1 second (FEV1) >= 50%
* Forced vital capacity (FVC) >= 50%
* Negative pregnancy test performed =< 7 days prior to registration, for women of childbearing potential only
* Willing to return to Mayo Clinic Rochester, Mayo Clinic Arizona, Mayo Clinic Florida for treatment

  * Note: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide blood and bone marrow samples for correlative research purposes

Exclusion Criteria:

* Prior autologous or allogeneic bone marrow/peripheral blood stem cell transplant
* More than two prior regimens for therapy of MM
* Myocardial infarction within 6 months prior to enrollment, or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; NOTE: Prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Seroreactivity for human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV) I or II, hepatitis B virus (HBV), hepatitis C virus (HCV)
* Other active malignancy < 2 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Any of the following:

  * Pregnant women or women of reproductive capability who are unwilling to use effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 28 days after stopping treatment
* Other co-morbidity, which would interfere with patient's ability to participate in the trial, e.g. uncontrolled infection, uncompensated lung disease
* Concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Known allergies to any of the components of the investigational treatment regimen or required ancillary treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06-04 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hayman, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Dose Level 3; Phase 2: Dose Level 3: CONDITIONING: Patients receive 56 mg/m^2 carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive 100mg/m^2 melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
- Phase 1: Dose Level 2: CONDITIONING: Patients receive 45 mg/m^2 carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive 100mg/m^2 melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
- Phase 1: Dose Level 1: CONDITIONING: Patients receive 36 mg/m^2 carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive 100mg/m^2 melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
- Phase 1: Dose Level 0: CONDITIONING: Patients receive 27 mg/m^2 carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive 100mg/m^2 melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
Period: Overall Study
Arm/Group | Phase 1: Dose Level 3 | Phase 1: Dose Level 2 | Phase 1: Dose Level 1 | Phase 1: Dose Level 0 | Phase 2: Dose Level 3
Started | 6 | 3 | 3 | 2 | 36
Completed | 6 | 3 | 3 | 2 | 35
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients that began treatment
Groups:
- Phase 1; Dose Level 3; Phase 1; Dose Level 2; Phase 1; Dose Level 1; Phase 1; Dose Level 0; Phase 2: CONDITIONING: Patients receive carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase 1; Dose Level 3 | Phase 1; Dose Level 2 | Phase 1; Dose Level 1 | Phase 1; Dose Level 0 | Phase 2 | Total
Number analyzed (Participants) | 6 | 3 | 3 | 2 | 35 | 49
Age, Continuous [Median (Full Range); unit: years] | 52 [42 to 65] | 61 [44 to 63] | 61 [60 to 66] | 55 [50 to 60] | 61 [46 to 77] | 60 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 14 | 17
  Male | 4 | 2 | 3 | 2 | 21 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 3 | 2 | 2 | 32 | 45
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose by the Number of Patients With a DLT Per Dose Level
Description: Will be defined as the dose level below the lowest dose that induces dose-limiting toxicity(DLT) in at least one-third of patients. For this study, a DLT is any of the following during the first 2 cycles of treatment; Absolute neutrophil count engraftment* delayed beyond day 21 or Platelet engraftment* delayed beyond day 30, grade 3+ related sensory or motor neuropathy, or grade 4+ related non-neurologic or non-hematologic adverse event(excluding nausea, vomiting, and diarrhea. Reported below are the number of patients who experienced a DLT.
Time Frame: Up to day 30
Population: All phase 1 patients that began treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Level 3 | Phase 1: Dose Level 2 | Phase 1: Dose Level 1 | Phase 1: Dose Level 0
Number analyzed (Participants) | 6 | 3 | 3 | 2
Participants | 1 | 0 | 0 | 0

2. Primary Outcome: Percentage of Patients With Complete Responses, Defined as a Complete Response Noted as the Objective Status on Two Consecutive Evaluations (Phase II)
Description: The percentage of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success percentages will be calculated.
Time Frame: Up to 5 years
Population: All patients that received dose level 3 treatment, including phase 1: dose level 3 patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Dose Level 3: CONDITIONING: Patients receive 56 mg/m^2 carfilzomib IV over 30 minutes on days -6, -5, -2, and -1. Patients also receive melphalan IV over 1 hour on days -4 and -3. TRANSPLANT: Patients undergo autologous stem cell transplant on day 0. Autologous Bone Marrow Transplantation: Undergo autologous stem cell transplant. Autologous Hematopoietic Stem Cell. Transplantation: Undergo autologous stem cell transplant, Carfilzomib: Given IV. Laboratory Biomarker Analysis: Correlative studies, Melphalan: Given IV
Arm/Group | Dose Level 3
Number analyzed (Participants) | 41
percentage of patients | 21.95 [10.56 to 37.61]

3. Secondary Outcome: Adverse Event Rate, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: These results are reported in the adverse events section. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 5 years
Population: All patients that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Level 3 | Phase 1: Dose Level 2 | Phase 1: Dose Level 1 | Phase 1: Dose Level 0 | Phase 2: Dose Level 3
Number analyzed (Participants) | 6 | 3 | 3 | 2 | 35
Participants | 6 | 3 | 3 | 2 | 35

4. Secondary Outcome: Complete Response Rate at Day 100
Description: Complete response rate (CRR) is defined as the percentage of complete responses estimated by the total number of patients who achieve a complete response by day 100 post-transplant divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true complete response rate at day 100 will be calculated.
Time Frame: At day 100
Population: All patients treated at dose level 3
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Level 3
Number analyzed (Participants) | 41
percentage of patients | 17.07 [7.15 to 32.06]

5. Secondary Outcome: Progression Free Percentage at 1 and 2 Years Post Registration
Description: Progression is an Increase of 25% from lowest value in any of the following (A "25% increase" refers to M protein, FLC and bone marrow results and does not refer to bone lesions, soft tissue plasmacytoma or hypercalcemia. The lowest value does not need to be a confirmed value. If the lowest serum Mprotein is ≥ 5 g/dL, an increase in serum M-protein of ≥ 1 g/dL is sufficient to define disease progression.), (In the case where a value is felt to be a spurious result per physician discretion (for example, a possible lab error), that value will not be considered when determining the lowest value.): Serum M-protein (absolute increase must be ≥ 0.5 g/dL) and/or Urine M-protein (absolute increase must be ≥ 200 mg/24 hrs) and/or If the only measurable disease is FLC, the difference between involved and uninvolved FLC levels (absolute increase must be>10 mg/dL) and/or If the only measurable disease is BM, bone marrow PC percentage (absolute increase must be ≥ 10%) (Bone marrow criteria for PD
Time Frame: At 1 year and 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Level 3
Number analyzed (Participants) | 41
percentage of patients
  1 year | 90.24 [76.87 to 97.28]
  2 years | 75.61 [59.70 to 87.64]

ADVERSE EVENTS:
Time Frame: 5 years
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s). The maximum grade for each type of adverse event will be recorded for each patient.
Arm/Group | Phase 1; Dose Level 3 | Phase 1; Dose Level 2 | Phase 1; Dose Level 1 | Phase 1; Dose Level 0 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/2 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/3 | 1/3 | 2/2 | 16/35
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 2/2 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Dose Level 3 (N=6) | Phase 1; Dose Level 2 (N=3) | Phase 1; Dose Level 1 (N=3) | Phase 1; Dose Level 0 (N=2) | Phase 2 (N=35)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Dose Level 3 (N=6) | Phase 1; Dose Level 2 (N=3) | Phase 1; Dose Level 1 (N=3) | Phase 1; Dose Level 0 (N=2) | Phase 2 (N=35)
Anemia (Blood and lymphatic system disorders) | 6 (9) | 2 (2) | 3 (3) | 2 (3) | 31 (45)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 8 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (8)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 15 (21)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 4 (5) | 2 (4) | 1 (2) | 0 (0) | 14 (25)
Lymphocyte count decreased (Investigations) | 4 (7) | 3 (6) | 3 (6) | 2 (4) | 32 (76)
Neutrophil count decreased (Investigations) | 5 (6) | 3 (11) | 3 (3) | 2 (3) | 30 (66)
Platelet count decreased (Investigations) | 6 (14) | 3 (13) | 3 (8) | 2 (4) | 35 (100)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 6 (11) | 3 (12) | 3 (4) | 2 (3) | 32 (82)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (10)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 12 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 4 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (10) | 2 (4) | 2 (7) | 2 (8) | 19 (52)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (18)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT01842308/Prot_SAP_000.pdf